CLINICAL TRIAL: NCT03751345
Title: Integrating Computer-Assisted Parent Training Therapy Into Community Mental Health Clinic Practice
Brief Title: Computerized Parenting Intervention
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rhode Island Hospital (Other)
Responsible Party: Principal Investigator, Jennifer Wolff, Staff Psychologist, Rhode Island Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1R34MH113598-01A1 (NIH)
Record Dates: First submitted 2018-10-02; First posted 2018-11-23 (Actual); Last update posted 2018-11-23 (Actual); Status verified 2018-11

CONDITIONS: Parenting; Adolescent Problem Behavior
Keywords: Parenting skills; Computer-based parenting program; Parenting Wisely; Adolescent disruptive behavior disorders

STUDY DESIGN:
Intervention Model Description: In the Open Trial, all participants will receive PW. In the RCT phase, adolescents will be randomly assigned to one of the two conditions. After completion of the baseline assessment, random assignment of adolescents using blocking and stratification will be automatically generated by the electronic data capture software REDCap. Random block sizes of assignments will be generated to prevent guessing of pending treatment assignments. Stratification will be used to ensure a balance on biological sex and disruptive behavior disorder severity (more of less than T=85), as indicated on the CBCL.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment As Usual (TAU) (No Intervention): The TAU condition consists of the standard treatment elements offered to all Gateway (study site) patients, and will be received by patients in both the PW and the TAU-only condition. TAU services during the adolescent's treatment are typically eclectic and mainly entail meeting with the adolescent alone to provide support and psychoeducation, with occasional family therapy sessions. Medication management is offered as needed.
- Parenting Wisely (PW) (Experimental): In addition to TAU services, the PW arm includes in-person sessions where parents complete computer-administered PW sessions, in-person session including therapist coaching to reinforce PW material and personalize treatment by applying PW skills to individual issues, and access to PW material remotely so parents can access information and skills from home as needed.
  Interventions: Behavioral: Parenting Wisely

INTERVENTIONS:
Behavioral: Parenting Wisely — PW is a self-administered, interactive, multimedia online program. Parents will complete computer-administered sessions during in-person appointments.The program comes with a parent workbook so that parents can gain additional exposure to and practice with the skills. The complete PW program takes from 3 to 5 hours to complete depending on the users' speed and depth of use. Parents will be given a login at enrollment so that they have the option to practice sessions or view any additional sessions at home. Individual coaching sessions will take place in-person with parents. Coaching sessions are designed to tailor the PW skills to each parent's presenting concerns.
  Other Names: PW
  Arms: Parenting Wisely (PW)

SUMMARY:
This study will evaluate a low-cost, low-intensity, computer-based model for delivering parenting skills to parents of adolescents in a community mental health clinic. This intervention has the potential to improve public health and community practice by making empirically-supported treatment techniques more available. We believe this approach will improve the efficiency of treatment delivery by integrating computerized and therapist delivered approaches, and there is potential for significant improvements in efficacy of parent training with this model.

DETAILED DESCRIPTION:
This study will evaluate a low cost, low intensity, technology based model for delivering parenting skills to parents of adolescents in a community mental health clinic (CMHC). Specifically, we will test a computer-assisted protocol of Parenting Wisely, a computer based parenting program with previously established efficacy. Such an intervention is consistent with NIMH strategic plan objective 3.3: "to strengthen the application of mental health interventions in diverse care settings by examining community and intervention delivery approaches and how they may affect intervention outcomes." Although this is a pilot effectiveness study, we will gather information to inform future implementation efforts including the feasibility and acceptability of the intervention. Additionally, we will conduct qualitative interviews with relevant stakeholders (providers/program managers) to better understand barriers and facilitators of adoption and sustainability. This goal will help increase the likelihood of a successful, future larger trial across multiple CMHCs due to its focus on external validity and implementation barriers when making critical design decisions. This approach mitigates a major criticism of traditional efficacy/effectiveness studies, i.e. that the methods do not translate well to the community due to cost and resource constraints, as well as contextual factors.

The intervention has the potential to improve public health and community practice by making empirically supported treatment techniques more available in CMHCs and improving the efficiency of treatment delivery by integrating computerized and therapist delivered approaches. Specifically, this study has the potential to advance treatment by: 1) understanding factors that enhance or impede computer assisted parent training in the community setting; 2) addressing a high-needs underserved population with significant public health relevance; 3) engaging the target mechanism of therapist fidelity, competency, and alliance as well as parenting skills and self-efficacy that have been shown to influence adolescent behavior problems; 4) increasing access to and engagement in an evidence-based treatment that can be personalized to the specific parenting skills of a family by the selection of modules in PW; and 5) enhancing the ease of dissemination and implementation. Furthermore, we believe this approach has the potential for improving response rate, because the parenting skills will be delivered with greater fidelity than would be typical of therapists teaching parenting in sessions in CHMCs. This improvement should also result in an improved response in adolescent behavior. We believe this is true because: 1) meta-analyses typically report moderate effect sizes for parent training at the end of treatment; 2) parent training is underemployed in community clinics; 3) fidelity to treatment protocols is often poor which has been shown to diminish effectiveness of treatment; and 4) frequent staff turnover creates high resource demands. Thus, we believe this approach is not only efficient but that there is potential for significant improvements in efficacy of parent training with this model.

ELIGIBILITY:
Inclusion Criteria:

* be the parent or legal guardian of an adolescent aged 12-17 years
* have an adolescent with clinically elevated disruptive behaviors as indicated by parent report on the Child Behavior Checklist (CBCL; Achenbach, 2000; Aggressive Problems or Oppositional/Defiant Problems T score > 70)
* be willing to receive a parenting intervention
* be fluent in English or Spanish
* be willing to provide written consent and teen willing to provide written assent

Exclusion Criteria:

* severe clinical presentations, such as psychosis or developmental delay, at a level that would interfere with the ability to assent or complete assessments

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2018-10-29 (Actual); Primary Completion 2021-05 (Estimated); Study Completion 2021-05 (Estimated)

PRIMARY OUTCOMES:
Change in Psychometric Analysis of the Perceptions of Computerized Therapy Questionnaire-Patient Version | Change from Baseline Psychometric Analysis of the Perceptions of Computerized Therapy at 6 months
  The PCTQ-P is an instrument for assessing consumers' perceptions of computer-based therapies that are distinguishable from traditional help-seeking attitudes. There are 35 items that can be divided in 6 sub-scales to measure subtle perceptions; relative advantage, compatibility, complexity, observability, trial-ability and future use intentions.
Consumer Satisfaction Questionnaire | 3 months after start of intervention
  The CSQ asks parents to rate their satisfaction with treatment delivery, their child's treatment progress, and their ability to manage their child's problems. Parents rate 11 items along a 7-point scale and answer 5 open-ended questions about their experience in treatment
Change in Psychometric Analysis of the Perceptions of Computerized Therapy Questionnaire- Clinician Version | Change from Baseline Psychometric Analysis of the Perceptions of Computerized Therapy at 3 months and 6 months
  an instrument for assessing clinicians' perceptions of computer-based therapies that are distinguishable from traditional help-seeking attitudes. There are 35 items that can be divided in 6 subscales to measure subtle perceptions; relative advantage, compatibility, complexity, observability, trial-ability and future use intentions.
Change in Evidence-Based Practice Attitude Scale | Change from Baseline Evidence-Based Practice Attitude Scale at 3 months and 6 months
  A 15 question reliable tool to evaluate the attitudes of providers who specialize in child and adolescent mental health toward Evidence Based Practice.
Change in Perceived Characteristics of Intervention Scale | Change from Baseline Perceived Characteristics of Intervention Scale at 3 months and 6 months
  The PCIS is a 20 question reliable assessment measure of perceived characteristics of interventions, and will be specified towards the intervention, Parenting Wisely.
Change in Qualitative Interviews | Change from Baseline Qualitative Interviews at 3 months and 6 months
  Qualitative feedback from interviews with parents, providers, and program managers will also be conducted. All quaAlitative interviews will be videotaped, transcribed verbatim and coded for nonverbal behaviors in addition to verbal content. We will use an interview guide to ensure the adequacy and quality of data. The guide will be refined to reflect unanticipated topics that arise and integrate these emergent topics and questions[40]. We will approach the interview as a collaborative process with participants and interviewers will encourage each participant to talk freely about the therapeutic process, coverage of parenting skills, and topic areas in PW. Broad questions will be followed by probes and unstructured questions based on areas raised by participants to encourage elaboration and clarification but limit influence from the interviewer.
Change in Pediatric Symptom Checklist | Change from Screening Pediatric Symptom Checklist at 3 months and 6 months
  A well-known measure to help primary care providers assess the likelihood of finding any mental health disorder in their patient. The questionnaire consists of 17 items on behavior or emotional problems.

SECONDARY OUTCOMES:
Parent Monitoring Questionnaire | Baseline assessment, 3 months after start of intervention, 6 months after start of intervention
  The PMQ is a 24 item youth and parent report measure designed to assess parental monitoring and sources of parental knowledge. The monitoring subscale has demonstrated good reliability (alpha = .82 parents, .85 youth) and correlates with adolescent internalizing and externalizing maladjustment, deviant peer relationships, and family discord.
McMaster Family Assessment Device | Baseline assessment, 3 months after start of intervention, 6 months after start of intervention
  This measure includes the following sub-scales assessing parenting skills: Problem Solving (i.e., the family's ability to resolve problems in ways that maintain effective family functioning.); Family Roles (i.e., the extent to which tasks are clearly and equitably distributed among family members); Communication (i.e., the extent to which verbal messages between family members are clear); Affective Involvement (i.e., the extent to which family members are interested in and placed value on each other's activities); Affective Responsiveness (i.e., the extent to which family members experience appropriate affect in response to stimuli); Behavioral Control (i.e., the extent to which the family expresses and maintains standards for the behavior of its members). All items are rated on a 4-point scale and the sub-scales have adequate reliability.
Parent-Adolescent Communication Scale | Baseline assessment, 3 months after start of intervention, 6 months after start of intervention
  The PACS is a youth and parent report measure that assesses positive and negative aspects of general parent-teen communication and the content and process of parent-teen interactions. The two sub-scales have good reliability (alpha = .77 - .88) and have been shown to correlate with teen engagement in problem behavior.
Parenting Self Efficacy | Baseline assessment, 3 months after start of intervention, 6 months after start of intervention
  This 10-item scale assesses the degree of parents' confidence in implementing specific parenting skills.
FAsTask Video Code | Baseline assessment, 3 months after start of intervention, 6 months after start of intervention
  The FAsTask is a video-taped family problem solving task that will be used to provide an in-vivo assessment of parenting behaviors. We have limited the assessment to tasks that align with our primary aims. Specifically, parent-teen dyads will be prompted to spend 5 minutes on each of the following: 1) teen leads a discussion about a time without supervision and parents seek additional information (monitoring and listening); 2) parents lead a discussion on setting limits over the previous month (limit setting) and then communicate rules to the teen; 3) parents and teens problem solve around an issue; and 4) positive recognition when the parent praises the teen.
Issues Checklist | Baseline assessment, 3 months after start of intervention, 6 months after start of intervention
  This measure will work to decipher distressed families versus non distressed families and addressing and identifying the issues.
Disruptive Behavior Disorder Rating Scale | Baseline assessment, 3 months after start of intervention, 6 months after start of intervention
  The DBDRS which is comprised of the DSM symptom lists for ADHD, ODD, and CD. It uses a 4-point response scale completed by parents for questions regarding ADHD and ODD and a yes/no format for CD symptoms to assess behavior problems within the past month. The DBDRS has been shown to have excellent psychometric properties
Child and Adolescent Services Assessment (CASA) | Baseline assessment, 3 months after start of intervention, 6 months after start of intervention
  This is a semi structured interview for parents and teens/children to assess service utilization for emotional, behavioral, and substance use problems. It addresses a range of services including inpatient, emergency room services, residential treatment centers, detention centers, probation, foster home services, hospitalization, in-home services, family therapy and outpatient services. The teen will complete questions regarding services related to school including boarding school, therapeutic/behavioral school, school support and school professional services
Working Alliance Inventory | 3 months after start of intervention.
  The WAI is an 11-item measure in which parents are asked to rate their alliance with their therapists on a 7-point Likert scale. This measure examines factors such as having a collaborative approach to treatment, perceived expertise, trust, and establishing shared goals.

CONTACTS AND LOCATIONS:
Locations (1):
- Gateway Healthcare Inc, Pawtucket, Rhode Island, United States